CLINICAL TRIAL: NCT03235622
Title: Women Health Cohort for Breast, Bone and Coronary Artery Disease
Acronym: BBC
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jung-Won Suh, Professor, Seoul National University Hospital
Other Study IDs: B-1707-406-102
Record Dates: First submitted 2017-07-24; First posted 2017-08-01 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Mammography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Coronary CT angiography — Presence of coronary plaques Characteristic of coronary plaques
  Other Names: Bone DEXA; Mammography

SUMMARY:
A single center cohort which enrolled women who performed mammography, bone densitometry (DEXA), and coronary CT angiography in Seoul National University Bundang Hospital from March 2011 to February 2013.

DETAILED DESCRIPTION:
To evaluate whether bone mineral density and breast arterial calcification can predict coronary artery disease in women older than 40 years

ELIGIBILITY:
Inclusion Criteria:

* Women (≥ 40 years) who performed mammography, bone DEXA, and coronary CT angiography at health promotion center of Seoul National University Bundang Hospital.

Exclusion Criteria:

* Women who have history of breast surgery or intervention
* Women who have history of myocardial infarction or revascularization
* Too poor image quality of coronary CT angiography for interpretation
* Renal dysfunction with serum creatinine ≥ 1.4mg/dL

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * The number of women who met inclusion criteria was 2113.
  * 13 women were excluded due to history of coronary revascularization (n=1) and breast surgery or intervention (n=12).
  * Finally, 2100 women were enrolled to the BBC cohort.
Sampling Method: Non-Probability Sample
Enrollment: 2100 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Presence of coronary plaque | 5 years
  Any coronary plaque in coronary CT angiography

SECONDARY OUTCOMES:
Characteristics of coronary plaque | 5 years
  Plaque characteristics (fibrosis, calcification, lipid, thrombosis) in coronary CT angiography
Major adverse cardiovascular events | 5 years
  Cardiac death, nonfatal myocardial infarction, ischemic stroke, coronary revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Won Suh, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yoon YE, Kim KM, Han JS, Kang SH, Chun EJ, Ahn S, Kim SM, Choi SI, Yun B, Suh JW. Prediction of Subclinical Coronary Artery Disease With Breast Arterial Calcification and Low Bone Mass in Asymptomatic Women: Registry for the Women Health Cohort for the BBC Study. JACC Cardiovasc Imaging. 2019 Jul;12(7 Pt 1):1202-1211. doi: 10.1016/j.jcmg.2018.07.004. Epub 2018 Aug 15. PMID 30121271